CLINICAL TRIAL: NCT07391332
Title: Psilocybin AsSisted pSychotherapy for the treatmENt of Gambling disordER : a Pilot Study
Acronym: PASSENGER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC25_0105; 2025-522743-18-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychotherapy assisted by high-dose psilocybin (25mg or 40mg where appropriate) (Experimental)
  Interventions: Drug: Psychotherapy assisted by high-dose psilocybin (25mg or 40mg where appropriate)
- Psychotherapy assisted by low-dose psilocybin (1 mg) (Active Comparator)
  Interventions: Drug: Psychotherapy assisted by low-dose psilocybin (1 mg)

INTERVENTIONS:
Drug: Psychotherapy assisted by high-dose psilocybin (25mg or 40mg where appropriate) — The first session of psilocybin PEX010 administration will use a moderately high dose of psilocybin, i.e., 25 mg. The dose may be increased to 40 mg during the second administration session in the experimental group, depending on the response during the previous session, as assessed by the Mystical Experience Questionnaire-30 (MEQ-30).
  Arms: Psychotherapy assisted by high-dose psilocybin (25mg or 40mg where appropriate)
Drug: Psychotherapy assisted by low-dose psilocybin (1 mg) — The first session of psilocybin PEX010 administration will use a very low dose of 1 mg in the control group. During the second administration session, the dose will be maintained at 1 mg.
  Arms: Psychotherapy assisted by low-dose psilocybin (1 mg)

SUMMARY:
The PASSENGER project aims to conduct a pilot feasibility study of the implementation of a randomized clinical trial on psilocybin-assisted psychotherapy for the treatment of gambling disorder. Feasibility will be assessed by estimating the ability to retain participants until the end of the protocol. Other objectives of the study will be to generate preliminary efficacy data, identify clinical factors potentially associated with the intensity of the psychedelic experience (which determines the expected therapeutic effect), and conduct a preliminary assessment of the safety of the treatment under study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older
* With a confirmed diagnosis of current gambling disorder (diagnostic criteria according to DSM-5), regardless of severity.
* Able to complete self-assessment questionnaires
* Willing to start addiction treatment, or for whom treatment already undertaken is not sufficient
* Willing to undergo a blood test and ECG
* Written and oral comprehension of French
* Having signed an informed consent form before any procedure under study
* Affiliated with a French social security system
* Women of childbearing age with a negative pregnancy test and highly effective contraception (according to version 1.2 of March 2024 of the CTCG recommendations in Appendix 7)
* Men of childbearing age using effective contraception (according to version 1.2 of March 2024 of the CTCG recommendations).
* Negative result on urinary toxicology screening
* In the case of psychotropic treatment (excluding nicotine replacement therapy): stabilization of dosage or initiation for more than 1 month.

Exclusion Criteria:

* Medical conditions that would prevent safe participation in the trial (epilepsy, significantly impaired liver function (TP<50%), significantly impaired kidney function (GFR<90 mL/min), coronary artery disease, history of arrhythmia, heart failure, uncontrolled hypertension, history of stroke, severe asthma, hyperthyroidism, narrow-angle glaucoma, symptomatic prostatic hypertrophy, or bladder neck obstruction).
* Serious ECG abnormalities (including QTc prolongation = corrected QT)
* Current or past psychotic or bipolar disorder
* Other unstable psychiatric disorder
* Family history (first-degree relatives) of psychotic disorder or type 1 bipolar disorder
* Current high risk of suicide (according to the MINI 5.0 suicide risk module)
* History of hallucinogen use disorder or any use in the past year
* Current alcohol use disorder with a history of withdrawal symptoms
* Extreme thinness (BMI < 16.5) or obesity (BMI > 30)
* Major cognitive impairment (Mini-Mental State Examination score < 26)
* Allergy or hypersensitivity to psilocybin or any of the excipients contained in the investigational drug
* Taking UGT1A9, UGT1A10, ALDH, or ADH inhibitors
* Pregnancy or breastfeeding
* Current protective measures (guardianship and legal protection)
* Participation in another interventional research protocol involving another psychotherapeutic or pharmacological intervention that may have an impact on clinical progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Protocol completion rate | End of study (33 months)
  Proportion of randomized participants who completed all scheduled visits and procedures, including all PAP sessions/control sessions and follow-up assessments until the end of study participation.

SECONDARY OUTCOMES:
Feasibility of recruitment and the proposed experimental protocol. | End of study (33 months)
  Goal of recruiting 30 participants within the planned inclusion period achieved
Assessement of the acceptability of the proposed experimental treatment by patients and caregivers. | Month 1
  Self-reported acceptability by patients and caregivers
Assessment of personal self-efficacy (General Self-Efficacy Scale: GSES) | Month 1
  Changes in each arm, between baseline assessment (V0) and post-treatment assessment (V1) of personal self-efficacy (General Self-Efficacy Scale: GSES)
Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score, and the WHOQOL-SRPB spirituality score | Month 1
  Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score obtained post-administration, and the spirituality WHOQOL-SRPB at baseline
Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score, and the Self-Compassion Scale | Month 1
  Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score obtained post-administration, and the self-compassion score (Self-Compassion Scale: SCS)
Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score, and treatment expectations (Credibility/Expectancy Questionnaire: CEQ) | Month 1
  Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score obtained post-administration, and treatment expectations based on the Credibility/Expectancy Questionnaire (CEQ)
Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score, and personal self-efficacy (General Self-Efficacy Scale: GSES) | Month 1
  Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score obtained post-administration, and the personal self-efficacy based on General Self-Efficacy Scale (GSES)
Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score, and average dose of psilocybin administered during the two sessions | Month 1
  Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score obtained post-administration, and average dose of psilocybin administered during the two sessions
Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score, and measurement of blind maintenance | Month 1
  Correlation between the intensity of the psychedelic experience, measured by the Mystical Experience Questionnaire (MEQ-30) score obtained post-administration, and the measurement of blind maintenance.
Clinical global impression of severity (Clinical Global Impression-Severity: CGI-S) | Month 1
  Changes between baseline assessment (Visit 0) and post-treatment assessment (Visit 1) of clinical global impression of severity (Clinical Global Impression-Severity: CGI-S)
Self-Compassion Scale (SCS) | Month 1
  Changes between baseline assessment (Visit 0) and post-treatment assessment (Visit 1) of Self-Compassion Scale (SCS)
Spirituality assessment (World Health Organization Quality of Life Spirituality, Religiousness and Personal Beliefs Instrument: WHOQOL-SRPB) | Month 1
  Changes between baseline assessment (Visit 0) and post-treatment assessment (Visit 1) of World Health Organization Quality of Life Spirituality, Religiousness and Personal Beliefs Instrument (WHOQOL-SRPB)
Analysis of daily diary | Month 1
  Changes between baseline assessment (Visit 0) and post-treatment assessment (Visit 1) of gambling behavior using daily diary.
Heart rate | Month 1
  Average scores in each arm of heart rate assessed during administration sessions
Blood pressure | Month 1
  Average scores in each arm of blood pressure assessed during administration sessions
Expected acute effects assessment | Month 1
  Average scores in each arm of expected acute effects (17-item behavior and mood observation grid), assessed during administration sessions
Assessment of Adverse Effects | Month 3
  Assessment of AEs (excluding expected acute effects), assessed during administration sessions in particular, but also throughout the duration of participation in the study;
Mini International Neuropsychiatric Interview (MINI 5.0) | Month 3
  Average scores in each arm of an increase in the level of suicide risk assessed by the Mini International Neuropsychiatric Interview (MINI 5.0)
Clinical Global Impression-Efficacy Index: CGI-IE | Month 3
  Average scores in each arm of the therapeutic index (Clinical Global Impression-Efficacy Index: CGI-IE) and clinical improvement (Clinical Global Impression-Improvement: CGI-I), assessed at post-treatment evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No